CLINICAL TRIAL: NCT05770557
Title: Survey on Attitudes About COVID-19 Vaccinations in a Survey of Italian Healthcare Workers
Brief Title: Survey on Attitudes About COVID-19 Vaccinations in Italian HCW
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4104
Record Dates: First submitted 2023-03-13; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Vaccination Hesitancy
MeSH Terms: conditions — Vaccination Hesitancy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: survey — administration of a survey among healthcare workers

SUMMARY:
The Project is aimed at analyzing the perceptions, knowledge, attitudes and intentions of the population towards the anti-SARS-CoV-2 vaccine in order to identify the determinants of vaccine refusal/hesitancy, and to guide specific activities aimed at updating and the implementation of institutional communication strategies on the vaccine, involving health professionals and targeting the general population.

ELIGIBILITY:
Inclusion Criteria:

* healthcare workers residing in Italy

Exclusion Criteria:

* healthcare workers not residing in Italy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: healthcare workers residing in Italy, of any age and gender
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
KAB factors | 4 months
  Identify the factors associated with knowledge, attitudes and intentions towards the anti-SARS-CoV-2 vaccine and the appropriate vaccine hesitancy measurement tools based on the best scientific evidence for the construction of the survey questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli, Roma, RM, Italy